CLINICAL TRIAL: NCT00700960
Title: Observational Study on Efficacy on Glycaemic Control of Slow-acting Insulin Analogue in Type 2 Diabetes
Brief Title: Observational Study Describing Conditions for Administering Slow-acting Insulin Analogue With Oral Antidiabetic Agents in Type 2 Diabetes on Blood Glucose Control
Acronym: LIGHT
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-1859
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — initiation of an long acting insulin treatment in association with OAD at the discretion of the physician/diabetologist

SUMMARY:
This study is conducted in Europe. The aim of this observational study is to describe the conditions for the concomitant administration of a slow-acting insulin analogue with oral antidiabetics (OADs) in order to improve blood glucose control in type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* HbA1c level greater than 7% despite treatment with two (or three) oral antidiabetic drugs (OADs) at an optimal dose level
* Patient agreeing to take part in the study and capable of completing a self-questionnaire.

Exclusion Criteria:

* Hypersensitivity to insulin or to one of the excipients
* Treatment with insulin for at least 6 months
* Participant in a clinical trial for diabetes on entry into the observational study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 2745 (Actual)
Dates: Start 2007-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
HbA1c | After 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Paris La Défense, France

REFERENCES:
- [Result] Verges B, Brun JM, Tawil C, Alexandre B, Kerlan V. Strategies for insulin initiation: insights from the French LIGHT observational study. Diabetes Metab Res Rev. 2012 Jan;28(1):97-105. doi: 10.1002/dmrr.1288. PMID 22218757
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com